CLINICAL TRIAL: NCT06724757
Title: Survey for Caregivers Aged 50 and Over
Acronym: PPA
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal investigator, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Other Study IDs: 2025-2165
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Caregiver Wellbeing; Caregiver Mental Health; Caregivers; Health
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Caregiver: Caregivers aged 50 years old and older living in Quebec
  Interventions: Other: Health questionnaire

INTERVENTIONS:
Other: Health questionnaire — The intervention involves the completion and analysis of an online questionnaire designed to assess the health (mental, physical, social) of caregivers aged 50 and over in Quebec. This assessment is based on a combination of questionnaires (CARE, 4-item Zarit scale, 4-item GDS, 3-item UCLA loneliness scale, etc.).

SUMMARY:
There are more and more informal caregivers (PPA) in Quebec. Their increase between 2012 and 2018, according to data from the "General Social Survey - Care Given and Received," was significant, around 32%. The available data paint a typical portrait of a Quebec caregiver: (a) she is a woman, (b) aged between 50-55 years, (c) who devotes at least 3 hours of her time per week, on a regular basis, (d) to caring for an elderly parent. To this date, there is no reliable data on the health status-whether mental, physical, or social-of caregivers in Quebec. Yet this information is crucial because it affects the ability of caregivers to fulfill their role and, consequently, the stable health of the individuals they care for, allowing them to continue living at home. This situation exposes caregivers to a decline in their own health, and by extension, the health of those they care for. The fact that the typical Quebec caregiver is 50 years old or older increases the risk of health deterioration within the caregiver-care receiver pair. Indeed, age 50 is when the effects of physiological and pathological aging begin to impact the physical capacities of the elderly. Developing new practices that focus on the health characteristics of both caregivers and care receivers, in order to prevent health deterioration, is therefore a crucial step in supporting caregivers in their role and ensuring that care receivers can stay at home in good conditions for as long as possible.

The issue of caregivers' health is still under-addressed in Quebec, both in the scientific literature and in population surveys. It seems that caregivers need a comprehensive evaluation of their health status (physical, mental, and social), given the significant impact caregiving has on their health. Research conducted within the Living Lab, led by Dr. Beauchet's team, has helped develop tools and questionnaires that effectively assess the frailty of individuals aged 50 and over and produce reports that raise awareness about their health status, enabling them to implement future care solutions that meet their needs.

The overall objective is to assess the health status (mental, physical, social) of caregivers aged 50 and over, living in Quebec-through self-assessment to make them aware of their actual health condition and engage them in a process of self-care.

ELIGIBILITY:
Inclusion Criteria:

* Be a caregiver
* Be 50 years old or older
* Reside in Quebec for at least 6 months and 1 day of the year
* Have an internet connection with an electronic device (computer, touch tablet or smartphone)
* Read and understand written French or English. The questionnaire is only available in these 2 languages.

Exclusion Criteria:

* Living in a Centre d'Hébergement et de Soins de Longue Durée (CHSLD) (long-term care centre) or in the medicalized sector of a seniors' residence.
* Participate in a concurrent interventional study (study involving medication or therapeutic intervention, etc.).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers aged 50 years old and older living in Quebec
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Physical health using the CARE frailty scale | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  CARE is a frailty scale. The AgeTeQ team has developed this scale, which enables frailty to be assessed via a standardized self-questionnaire comprising 22 simple questions, 20 of which are based on a binary response (yes versus no) and two on numerical. CARE is based on a cumulative deficit approach to measuring frailty. Each response is assigned a point 1 if there is a deficit, and 0 if there is no deficit.
  The CARE score ranges from 0 (no deficits) to 21 (maximum cumulative deficits). This score has been segmented into 3 levels using a validated approach to determine 3 levels of frailty:
  * The robust level: score between 0 and 1.
  * Pre-fragile level: score between 2 and 4.
  * Fragile level: score > 5.

SECONDARY OUTCOMES:
Caregiver burden with the 4-item Zarit score (/20) | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  The caregiver burden is assessed using the 4-item Zarit scale. This scale asks four questions that reflect how caregivers feel when caring for their loved ones. For each statement, the respondent is asked to indicate a frequency: never, rarely, sometimes, quite often and almost always.
Depression with the 4-item GDS score (/4) | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  The Geriatric Depression Scale or GDS was designed to assess the presence of depressive feelings and suicidal intentions in the elderly. It is essentially a screening test for depressive impairment or state. The GDS is initially composed of 30 questions with a binary response choice (yes or no). For reasons of questionnaire length, it was decided to use an abbreviated version of the GDS with 4 items. The GDS then gives a score between 0 and 4, with 0 corresponding to a very high probability of no depression, and 1 or more corresponding to a very high probability of depression.
Social isolation | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  A question is asked to measure the social isolation of caregivers, taking into account the number of contacts (in person or by telephone) with people outside the household (friends, family, professionals).
Loneliness with the UCLA score (/9) | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  The 3-item UCLA scale is a screening tool for loneliness in adults. The scale consists of three questions, with frequency options: never, sometimes and often. The score can vary between 3 and 9. A high score indicates a high degree of loneliness.
Perceived health scores | Questionnaire completed once (15 minutes) between October 2024 and February 2025
  Three additional questions are asked in the form of a scale (ranging from 0 to 10) to assess the perceived health of caregivers. For each domain, the respondent is asked to indicate his or her state of perceived health, ranging from 0 (the worst state of health the respondent can imagine) to 10 (the best state of health the respondent can imagine). Three health domains are investigated: psychological health, physical health and social isolation.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided